CLINICAL TRIAL: NCT04775979
Title: Efficacy and Safety of Diphenylcyclopropenone (DPCP) as a Depigmenting Therapy in Extensive Vitiligo
Brief Title: Diphenylcyclopropenone (DPCP) as a Depigmenting Therapy in Extensive Vitiligo
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mayson, Resident, Ain Shams University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASUMS730/2020/2021
Record Dates: First submitted 2021-02-20; First posted 2021-03-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo | interventions — diphenylcyclopropenone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diphenylcyclopropenone (DPCP) (Experimental): Applying DPCP topically
  Interventions: Drug: diphenylcyclopropenone (DPCP)

INTERVENTIONS:
Drug: diphenylcyclopropenone (DPCP) — Depigmenting agent

SUMMARY:
The aim of the present work is to evaluate the efficacy and safety of diphenylcyclopropenone (DPCP) as a depigmenting therapy in extensive Vitiligo.

DETAILED DESCRIPTION:
Depigmentation protocol: (Aghaei et al, 2005)

* Substance used: DPCP (FLUKA, Sigma-Aldrich, Saint Louis, MO (Missouri), USA) 98% pure powder.
* DPCP will be dissolved in acetone to obtain 2% solution.
* DPCP solutions will be kept in dark colored bottles at 4ºC (degree Celsius).
* Sequential dilution by acetone to yield 1%, 0.5%, 0.1%, 0.01%, 0.05 and 0.001%.
* Sensitization by DPCP concentration 2% will be applied to an area 5×5 cm on the forearm
* Two weeks following sensitization, treatment will be started by weekly applications of incremental concentrations of DPCP (between 0.001% and 2%) adjusted according to the patient's reactivity to the contact allergen. The aim will be to maintain mild contact eczema and itch for about 48 hours after application. Patients will be instructed to avoid direct sun exposure of the treated area and not to wash it for 48 hours after each application.

Patient follow-up: Patients will come for sensitization at week 0, then after 2 weeks to look for the allergic response, then weekly to reach the effective dose of DPCP. After reaching the effective dose, patients will come weekly to apply DPCP and to look for depigmentation, record possible side effects for 12 consecutive weeks.

Assessment of depigmentation:

For each treated area, response will be assessed as follows (van Geel et al., 2015):

* Digital clinical pictures will be used to evaluate the capacity to induce depigmentation and to assess the percentage of depigmentation per test area.
* Treatment results will be subsequently classified according to a grading system from 0 to 6 (0 = no effect, 1 = <25%; 2 = 25-49%; 3= 50-47%; 4= 50-74%; 5=90-99%; 6=100%), corresponding to the grade of depigmentation.

Reporting any side effects: such as pain, erythema, blisters, erosions, hyperpigmentation, scarring, appearance of depigmentation in distant sites and/or systemic manifestations (Venkatesh et al,2018) .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients of both genders ≥ 18 years.
2. Vitiligo universalis patients with cosmetically unacceptable residual pigmentation.
3. Extensive vitiligo vulgaris ≥ 50% body surface area (BSA) involvement with areas recalcitrant to repigmentation on exposed skin with consequent psychological impairment.

Exclusion Criteria:

1. Children.
2. Early, localized, segmental or any vitiligo case responsive to repigmentation treatment.
3. Pregnant and lactating females.
4. Patients with history of any malignancy.
5. Patients with active infectious or inflammatory dermatoses.
6. Patients with a history of hypertrophic scars or keloids.
7. Patients suffering from cardiac, hepatic or renal disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-17 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Depigmentation | 6 weeks
  Assessment of depigmentation:
  For each treated area, response will be assessed as follows (van Geel et al., 2015):
  * Digital clinical pictures will be used to evaluate the capacity to induce depigmentation and to assess the percentage of depigmentation per test area.
  * Treatment results will be subsequently classified according to a grading system from 0 to 6 (0 = no effect, 1 = <25%; 2 = 25-49%; 3= 50-47%; 4= 50-74%; 5=90-99%; 6=100%), corresponding to the grade of depigmentation.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa MA Abdallah, Study Chair — Ain Shams University; Rania M Elhusseiny, Study Director — Ain Shams University
Locations (1):
- University hospitals faculty of medicine ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No